CLINICAL TRIAL: NCT03109340
Title: Efficacy of Moderate Intensity Walking Provided Feedback by ECE PEDO on Abdominal Fat in Women With Overweight and Obesity
Brief Title: Efficacy of ECE PEDO (Equipment for Clever Exercise) on Abdominal Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Füsun Ardıç, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013TPF009
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Obesity, Abdominal; Physical Activity
Keywords: abdominal obesity; walking; aerobic exercise
MeSH Terms: conditions — Obesity, Abdominal; Motor Activity

STUDY DESIGN:
Intervention Model Description: Women with overweight and obesity were assigned to two groups: supervised treadmill walking (Group I) or walking with ECE PEDO (Group II).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised treadmill group (Active Comparator): a. Supervised treadmill group (Group I): The participants were instructed walking exercise at their target heart rate on a treadmill in Sports Rehabilitation Unit of Pamukkale University.
  Interventions: Other: Supervised treadmill group (Group I)
- ECE PEDO pedometer group (Experimental): b. ECE PEDO® pedometer group (Group II): Participants were given the walking program with ECE PEDO giving audible feedback in case of any deviation from their target range of steps per minute.
  Interventions: Device: ECE PEDO pedometer (Group II)

INTERVENTIONS:
Other: Supervised treadmill group (Group I) — An exercise prescription was developed for each woman on the basis of the data acquired from the baseline treadmill exercise test. Target HR corresponding to values of 50-70% VO2max (moderate-intensity) was determined by the submaximal treadmill test.The participants were instructed walking exercise at their target HR on a treadmill in Sports Rehabilitation Unit of Pamukkale University. HR was monitored by a Polar HR monitor (Polar Beat, Port Washington, NY).During 12 weeks, 5 days in a week and 30 minutes per day walking program was applied.
  Arms: Supervised treadmill group
Device: ECE PEDO pedometer (Group II) — Following a 10-minute rest after treadmill test, the participants were instructed to walk on the treadmill while maintaining their target heart rate. The number of steps taken in a minute was calculated using a criterion pedometer when target HR responses were reached. In this way, we determined the steps per minute required to moderate intensity walking for each participant. Detected individual step numbers were recorded to ECE PEDO for each person. Then participants were given the walking program with ECE PEDO giving audible feedback in case of any deviation from the range of steps per minute.During 12 weeks, 5 days in a week and 30 minutes per day walking program was applied.
  Arms: ECE PEDO pedometer group

SUMMARY:
Objective: To show the effectiveness of walking with ECE PEDO (Equipment for Clever Exercise) comparing supervised treadmill walking corresponding moderate aerobic exercise intensity on abdominal obesity and cardiorespiratory capacity.

DETAILED DESCRIPTION:
Objective: To show the effectiveness of walking with ECE PEDO (Equipment for Clever Exercise) comparing supervised treadmill walking corresponding moderate aerobic exercise intensity on abdominal obesity and cardiorespiratory capacity.

Methods: Twenty-eight women with overweight and obesity were assigned to two groups: supervised treadmill walking (Group I,n=14) or walking with ECE PEDO (Group II,n=14). Target heart rate(HR) corresponding to values of 50-70% VO2max were determined by the submaximal treadmill test. Group 1 was instructed walking at their target HR on a treadmill. The number of steps taken in a minute corresponding to target HR was determined by a criterion pedometer and group 2 was instructed walking in these step range recorded to ECE PEDO giving audible feedback. Before and after a 12-week exercise program, participants were evaluated by BMI and waist circumference(WC); ultrasonographic visceral fat thickness(VFT) and ergospirometric VO2max.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants who meet the criteria for inclusion were women with overweight weight or obesity and were 26-60 years old with a BMI (in kg/m2) from 27.1 to 39.6 and, waist circumference > 80 cm.

Exclusion Criteria:

* The exclusion criteria were BMI values less than 24.9 and higher than 40, presence of a atherosclerotic heart disease, musculoskeletal or systemic diseases contradicting the exercise, a neurological or psychiatric disease affecting cooperation and cognitive function, and participation in a calorie restricted diets.

Ages: 26 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 65 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2014-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in abdominal visceral fat thickness (VFT) at week 12. | Week 12.
  Ultrasonographic (US) imaging was performed by the convex probe with 3.5 Megahertz (General Electric Logic E9). Abdominal VFT measurement was done with the placement of probe transversely at 1 cm above of the umbilicus while the participant was lying in the supine position.
Change from baseline in body mass index (BMI) at week 12. | Week 12.
  Weight and height were measured with weight scale and stadiometer. Body mass index (BMI) was calculated for as weight (kg) divided by height squared (m2).
Change from baseline in waist circumference at week 12. | Week 12.
  Waist circumference was measured at the midpoint of the distance between the lowest rib and iliac crest with the non-elastic tape.

CONTACTS AND LOCATIONS:
Overall Officials: Fusun Ardic, Prof., Study Chair — University of Pamukkale

IPD SHARING:
Plan to Share IPD: Undecided
Plan not defined as work is completed